CLINICAL TRIAL: NCT05459259
Title: Development of an Optimal Physiotherapy Intervention for Arthrofibrosis Following Total Knee Replacement. ReSTART Study (Reducing Stiffness After Knee Replacement)
Brief Title: Physiotherapy for Arthrofibrosis Following Knee Replacement.
Acronym: ReSTART
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Collaborators: King's College London (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 22027
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Arthroplasty Complications; Fibrosis; Knee Joint Contracture
Keywords: knee stiffness
MeSH Terms: conditions — Fibrosis | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients participants: Adults who have undergone elective knee arthroplasty with post-operative arthrofibrosis/stiffness who have undergone MUA in the previous 24 months or are currently listed for a MUA.
  Interventions: Other: Interviews and Delphi Survey
- Healthcare Professionals: Physiotherapists/Occupational Therapist/ Nurses and Orthopedic surgeons with clinical experience in the management of patients with arthrofibrosis following knee joint arthroplasty
  Interventions: Other: Interviews and Delphi Survey

INTERVENTIONS:
Other: Interviews and Delphi Survey — no intervention delivered

SUMMARY:
This research aims to develop an optimal physiotherapy intervention for people with arthrofibrosis (stiffness due to scar tissue) after total knee replacement (TKR). We will develop an optimal intervention by conducting:

1. A review of the evidence to identify what components could be included in the intervention, how effective they are and what outcomes have been measured by the research.
2. Interviews with patients with arthrofibrosis to understand the impact it has on their life and what outcomes are important to them and interviews with healthcare professionals (HCPs) to understand their experiences of treating patients with arthrofibrosis.
3. A Delphi study with a larger group of HCPs and patients to reach a consensus on what the optimal intervention should include. This involves a series of anonymous voting on a range of items that have been generated by the group and the results of the evidence review.
4. A workshop with patients, HCPs and health-care commissioners to finalise the intervention. During the workshop we will present our findings and work in small groups to agree the intervention

ELIGIBILITY:
Inclusion Criteria for Patients:

* adults (aged 18 and over) of any age who have undergone elective TKR with post- operative arthrofibrosis/stiffness who have undergone manipulation under anaesthetic (MUA) in the previous 24 months or are currently listed for a MUA.
* Ability to give informed consent

Exclusion Criteria:

* Patients with neurological or blood disorders

For HCP participants :

* at least 5 years of experience working with joint arthroplasty including the management of patients with arthrofibrosis or 3 years in the case of orthopaedic surgeons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have had problematic stiffness following knee arthroplasty and healthcare professionals who manage patients with those conditions.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Qualitative interviews with Patients and Healthcare Professionals | 12 months
  we will conduct qualitative interviews with patients to explore (i) the experiences, important outcomes and unmet needs of patients; and with health care professionals (HCPs) to understand (ii) their experiences, perceptions and context of managing arthrofibrosis and (iii) their opinions on the intervention components identified in a systematic review of the evidence.
A Delphi survey with HCPs and patients to achieve consensus agreement on the most important components of an optimal intervention. | 6 months
  We will conduct a modified Delphi exercise with a maximum of 4 rounds to agree consensus on (i) the essential components of the intervention and what are the important outcomes that should be collected for patients with arthrofibrosis .

CONTACTS AND LOCATIONS:
Overall Officials: Michelle C Hall, PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moffatt F, Narayanasamy M, Smith B, Stock J, Sheehan K, Sackley C, Hall M. "My bloody leg" - The lived experience of arthrofibrosis after total knee arthroplasty. Physiotherapy. 2025 Oct 28;130:101862. doi: 10.1016/j.physio.2025.101862. Online ahead of print. PMID 41273943